CLINICAL TRIAL: NCT07326540
Title: A Phase 3 Prospective, Randomized, Multicenter, Active-controlled Study to Evaluate the Efficacy and Safety of BV100 Plus Low-dose Polymyxin B Compared With Colistin Plus High-dose Ampicillin/Sulbactam in the Treatment of Adult Patients With Hospital-acquired Bacterial Pneumonia and Ventilator-associated Bacterial Pneumonia Caused by Carbapenem-resistant Acinetobacter Baumannii-calcoaceticus Complex
Brief Title: Efficacy and Safety of BV100 Plus Low Dose Polymyxin B Versus Colistin Plus High-dose Ampicillin/Sulbactam in Patients With Hospital-acquired or Ventilator-associated Bacterial Pneumonia Due to Carbapenem-resistant Acinetobacter Baumannii-calcoaceticus Complex
Acronym: RIV-TARGET
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: BioVersys SAS (Industry)
Collaborators: BioVersys AG (Industry)
Responsible Party: Sponsor
Organization: BioVersys AG (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BV100-010
Record Dates: First submitted 2026-01-07; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Hospital Acquired Bacterial Pneumonia (HABP); Ventilator Associated Bacterial Pneumonia (VABP); Colistin Resistanrt ABC; Acinetobacter Baumannii-calcoaceticus Complex
Keywords: BV100; CRABC; VABP; HABP; polymyxin B; colistin
MeSH Terms: interventions — Polymyxin B; Colistin; sultamicillin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Part A - Group 1: BV100 (rifabutin for infusion) plus low dose polymyxin B (Experimental): Part A is the pivotal, assessor-blind, randomized, comparative portion of the study in patients with documented ABC hospital-acquired bacterial pneumonia (HABP) or ventilator-associated bacterial pneumonia (VABP).
  Part A - Group 1 (experimental): 300 mg BV100 plus 50 mg polymyxin B infused over 2 hours every 12 hours (q12h), plus 2 g meropenem infused over 1 hour every 8 hours (q8h)
  Interventions: Drug: BV100 (300 mg); Drug: Polymyxin B; Drug: MEROPENEM 2 grams TID
- Part A-Group 2: Colistin plus high dose ampicillin/sulbactam (Active Comparator): Part A - Group 1 (control group): Colistin (4,500,000 units intravenously [IV] over 1 hour q12h, after an initial loading dose of 9,000,000 units infused over 1 hour) plus high dose ampicillin/sulbactam (6 g/3 g IV over 4 hours q8h, plus 2 g meropenem infused over 1 hour every 8 hour (q8h).
  Interventions: Drug: Colistin; Drug: Ampicillin-Sulbactam; Drug: MEROPENEM 2 grams TID
- Part B-Group 3: BV100 (rifabutin for infusion) plus low dose polymyxin B (Experimental): Part B (Group 3) is the open-label, nonrandomized supportive portion of the study that includes patients known to have HABP or VABP associated with ABC organaisms resistant to colistin or polymyxin B, or who have who have failed a colistin or polymyxin B regimen prior to study entry. Part B - Group 3: 300 mg BV100 plus 50 mg polymyxin B infused over 2 hours every 12 hours (q12h), plus 2 g meropenem infused over 1 hour every 8 hours (q8h).
  Interventions: Drug: BV100 (300 mg); Drug: Polymyxin B; Drug: MEROPENEM 2 grams TID

INTERVENTIONS:
Drug: BV100 (300 mg) — 300 mg BV100 nfused over 2 hours every 12 hours (q12h).Treatment for 7 days up to 14 days if clinically indicated.
  Arms: Part A - Group 1: BV100 (rifabutin for infusion) plus low dose polymyxin B; Part B-Group 3: BV100 (rifabutin for infusion) plus low dose polymyxin B
Drug: Polymyxin B — 50 mg polymyxin B infused over 2 hours every 12 hours (q12h).Treatment for 7 days up to 14 days if clinically indicated.
  Arms: Part A - Group 1: BV100 (rifabutin for infusion) plus low dose polymyxin B; Part B-Group 3: BV100 (rifabutin for infusion) plus low dose polymyxin B
Drug: Colistin — Colistin (4,500,000 units infused over 1 hour every 12 hours (q12h), after an initial loading dose of 9,000,000 units infused over 1 hour).Treatment for 7 days up to 14 days if clinically indicated.
  Arms: Part A-Group 2: Colistin plus high dose ampicillin/sulbactam
Drug: Ampicillin-Sulbactam — High dose ampicillin/sulbactam (6 g/3 g IV over 4 hours q8h).Treatment for 7 days up to 14 days if clinically indicated.
  Arms: Part A-Group 2: Colistin plus high dose ampicillin/sulbactam
Drug: MEROPENEM 2 grams TID — meropenem infused over 1 hour every 8 hours (q8h).Treatment for 7 days up to 14 days if clinically indicated.

SUMMARY:
This is a two-part study, with Part A being the randomized, controlled portion of the study in patients with hospital-acquired bacterial pneumonia (HABP) or ventilator-associated bacterial pneumonia (VABP) suspected or confirmed to be due to carbapenem-resistant Acinetobacter baumannii-calcoaceticus complex (CRABC).

Part B is the single-group portion of the study and includes patients with HABP or VABP with CRABC infections that are resistant to or have failed colistin/polymyxin B treatment.

DETAILED DESCRIPTION:
This is a Phase 3, randomized, active-controlled two-part parallel-group study to evaluate the efficacy and safety of BV100 plus low-dose polymyxin B in patients with HABP or VABP suspected or confirmed to be due to CRABC infection. Eligible patients who provide informed consent will be enrolled in the study and will have pretreatment blood and infection site-specific samples collected and submitted to a local laboratory. The overall study design consists of two parts in which patients will be recruited in parallel.

Part A is the pivotal, randomized, comparative portion of the study, focusing on patients with suspected or confirmed CRABC HABP or VABP. Part A of the study will employ a partially blinded design. Site personnel directly involved in patient care and treatment administration will be unblinded to treatment assignment; however, access to treatment allocation information, including data potentially revealing assigned treatment arm, will be restricted for Sponsor study personnel. No personnel employed at the Sponsor will have access to the data, maintaining blinding for all Sponsor employees. Project management and oversight and medical query management will be conducted by unblinded external providers or vendors. The Central Adjudication Committee (CAC) will be the blinded assessor.

Part B is a prospective multicenter, open-label, nonrandomized, additional single group to evaluate the efficacy and safety of BV100 plus low-dose polymyxin B in patients with HABP or VABP due to CRABC known to be resistant to colistin or polymyxin B prior to study entry and patients where colistin or polymyxin B regimen has failed prior to study entry. Approximately 25 patients are expected to be enrolled in Part B. Patients randomized to either group of Part A cannot be transferred to Part B.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent prior to any study related procedures not part of normal medical care. If permitted by local country and institution-specific guidelines, surrogate consent/use of a legally authorized representative may be provided. Alternatively, the decision can be made according to the procedure permitted by local law and institutional Standard Operating Procedures. If a patient regains consciousness while in the study and, per the Investigator's judgment, the patient is able to read, assess, understand, and make his/her own decision to participate in the study, the patient may agree to continue participation. In such cases, the patient must be reconsented.
2. Male or female patients, ≥ 18 and ≤ 82 years of age at the time of signing informed consent.
3. A confirmed diagnosis of HABP or VABP requiring treatment with IV antibiotics in the judgment of the Investigator.
4. High probability of a pneumonia (HABP or VABP) due to ABC as a single pathogen, or member of a polymicrobial infection based on evidence from RDT from a sample collected within 48 hours prior to randomization, AND one of the following:

   1. Has received no more than 48 hours of potentially active antimicrobial treatment against CRABC prior to the first dose of study drug; OR
   2. Is clinically failing prior treatment regimens (i.e., clinical deterioration or failure to improve after at least 48 hours of antibiotic treatment).
5. An APACHE II < 30 or qSOFA score ≥ 2 at Screening.
6. Women of childbearing potential must have a negative highly sensitive urine or serum pregnancy test before randomization. Participating women of childbearing potential must be willing to consistently use one highly effective method of contraception from Screening until at least 30 days after administration of the last dose of study drug.
7. Diagnosed with HABP or VABP

Exclusion Criteria:

1. For Part A only, patients with an infection known to be resistant to colistin, with a known intolerance to polymyxins, or taking any drug that prevents them from receiving polymyxins.
2. Evidence of active concurrent pneumonia requiring additional antimicrobial treatment caused by, e.g., Streptococcus pneumoniae, Haemophilus influenzae, Staphylococcus aureus, Mycoplasma pneumoniae, Chlamydia pneumoniae, Legionella pneumophila, Pneumocystitis jiroveci, Aspergillus spp, respiratory syncytial virus, influenza and parainfluenza viruses, Middle East respiratory syndrome coronavirus, mycobacteria, mucormycosis.
3. Any of the following health conditions:

   1. Pulmonary disease that precludes evaluation of a therapeutic response.
   2. Pleural empyema (exception: acceptable if drainage occurs within 24 hours of Screening and patient is expected to be treated in ≤ 14 days).
   3. Solid organ transplant within 6 months prior to randomization.
   4. Evidence of deep seated infection, e.g., Gram-negative osteomyelitis, or meningitis requiring prolonged therapy.
   5. Acute infective endocarditis due to Gram-positive bacteria that requires urgent treatment/emergent indication of surgery, or patients in whom surgery is contraindicated due to prohibitive risk for surgery due to comorbidities.
   6. Surgical wound infections requiring further surgical management e.g., wound closure, drain removal.
   7. Peritonitis.
   8. Irremovable implantable device or line thought to be the source of the ABC infection.
   9. Known or suspected neuropathy or neuromuscular disease.
   10. Human immunodeficiency virus infection.
   11. Chronic immunosuppression due to drugs and/or underlying disease
4. Bronchial obstruction or a history of post obstructive pneumonia (this does not exclude patients with pneumonia who have an underlying chronic obstructive pulmonary disease).
5. Patients classified under futility of care, as determined by the medical team, indicating a lack of potential for benefit from intervention or patients who are permanent residents of long-term care facilities and have been assessed by the clinical team as receiving palliative or comfort-focused care.
6. Sustained shock with persisting hypotension requiring vasopressors to maintain mean arterial pressure ≥ 65 mmHg
7. Diagnosis of ventilator-associated tracheobronchitis.
8. Inability to provide proper respiratory specimens for culture.
9. Received more than 48 hours of potentially active treatment against CRABC prior to the first dose of study drug.
10. Known or suspected allergy to polymyxin, rifabutin, colistin, ampicillin/sulbactam, meropenem or their excipients.
11. Acute graft-versus-host disease (Grade ≥ 3).
12. Requirement for continuing treatment with probenecid, methotrexate, ganciclovir, valproic acid, or divalproex sodium during the study.
13. Requirement at the time of randomization for any reason, or likely to require during the patient's participation in the study (from randomization through the EoS Visit), for additional systemic Gram-negative antimicrobial therapy potentially active toward CRABC.
14. Expected survival < 72 hours or a Do Not Resuscitate Order.
15. Burns > 40% of total body surface area.
16. Presence of neutropenia (absolute neutrophil count < 1500/mm3) obtained from a local laboratory at Screening, or anticipated neutropenia with absolute neutrophil count < 1500 cells/mm3.
17. Severe renal disease defined as an estimated glomerular filtration rate (eGFR) as per Modification of Diet in Renal Disease (MDRD) formula (MDRD eGFR) < 30 mL/min/1.73 m2, or requirement for peritoneal dialysis, hemodialysis, hemofiltration, or a urine output < 20 mL/hour over a 24 hour period.
18. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3× upper limit of normal (ULN) AND total bilirubin > 2×ULN at Screening (using local laboratory values); or Child Pugh Class C in patients with chronic liver function impairment. Evidence of significant hepatic disease or dysfunction, including known acute viral hepatitis, hepatic cirrhosis, hepatic failure, chronic ascites, or hepatic encephalopathy.

    Note: Patients with AST or ALT up to 5×ULN are eligible if these elevations are acute and are documented as being directly related to the infectious process being treated.
19. Investigator's opinion of clinically significant ECG finding such as new ischemic changes, infarct, or ventricular arrhythmia with immediate potential for a fatal outcome, bradycardia not corrected by pacemaker or medication, or, prior to the current infection, a history of New York Heart Association Class IV cardiac failure defined as severe limitations - experiences symptoms even while at rest, mostly bedbound patients, within 1 year.
20. Abnormal QT interval corrected for heart rate by Fridericia formula (QTcF): > 500 ms confirmed with repeat ECG.
21. Stroke (ischemic or intracerebral hemorrhage) within 10 days prior to randomization or expected survival from stroke < 28 days or Glasgow Coma Scale score 3 with no hope of improvement.
22. Women who are pregnant or nursing.
23. Patients who are currently enrolled in or have not yet completed, in the last 30 days or 5 half lives, whichever is longer, another investigational device or drug study or those who are receiving other investigational agents.
24. Unable or not willing, in the opinion of the Investigator, to comply with all study protocol.

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2026-03-20 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with All-Cause Mortality in CRABC m-MITT Population | Day 28
  The primary efficacy endpoint for the study is 28-day all-cause mortality (ACM) in the CRABC Microbiological Modified Intention-to-Treat (CRABC m-MITT) population in Part A.

SECONDARY OUTCOMES:
Proportion of Patients with clinical cure at ToC in CRABC m-MITT Population | 7 days after end of treatment
  Clinical cure status (cure, failure, indeterminate) will be assessed at the ToC in CRABC m-MITT Population in Part A